CLINICAL TRIAL: NCT04654585
Title: Sevrage Tabagique à l'Aide Des Outils dédiés Selon la Préférence, un Essai randomisé contrôlé Pragmatique
Brief Title: Preference-based Tools for Smoking Cessation Among Disadvantaged Smokers, a Pragmatic Randomised Controlled Trial
Acronym: STOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société de Formation Thérapeutique du Généraliste - Recherche (Other)
Collaborators: National Cancer Institute, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Fabienne El-Khoury, Senior researcher, principal investigator, Institut National de la Santé Et de la Recherche Médicale, France
Organization: Société de Formation Thérapeutique du Généraliste (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STOP-001
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Smoking; Smoking Cessation
Keywords: Electronic Nicotine Delivery Systems; Tobacco Use Cessation Devices; Preference-based
MeSH Terms: conditions — Smoking; Smoking Cessation; Vaping | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The STOP intervention (Experimental): The stop intervention is a heath professional (medical doctor) led intervention assisting smokers with low socioeconomic position in their smoking cessation attempt. It consists of routine care and adapted advice supplemented with a free delivery of any or several type(s) of nicotine replacement therapy (NRT) (patches, inhalers, gum, tablets, etc.) and/or an e-cigarette + e-liquid. The delivery of those smoking aids is based on the smokers' preference and choice.
  Interventions: Other: The STOP intervention
- Standard Care (Active Comparator): Participants randomised to the standard care group will be given standard care in assisting their smoking cessation attempt, but without free delivery of NRT or e-cigarettes.
  Standard care includes motivational interviewing, advice to quit and prescription for NRTs. The number and online address of the French smoking cessation support helpline could also be provided. Health professionals will also be in position to prescribe NRT or other treatments (for example: Varenicline or Bupropion) which can help with smoking cessation, according to routine practice. The health professional could also give advice on e-cigarette use if he or she finds it suitable.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: The STOP intervention — The stop intervention is a heath professional (medical doctor) led intervention assisting smokers with low socioeconomic position in their smoking cessation attempt. It consists of routine care and adapted advice supplemented with a free delivery of any or several type(s) of nicotine replacement therapy (NRT) (patches, inhalers, gum, tablets, etc.) and/or an e-cigarette + e-liquid. The delivery of those smoking aids is based on the smokers' preference and choice.
  Arms: The STOP intervention
Other: Standard Care — Participants randomised to the standard care group will be given standard care in assisting their smoking cessation attempt, but without free delivery of NRT or e-cigarettes.
  Standard care includes motivational interviewing, advice to quit and prescription for NRTs. The number and online address of the French smoking cessation support helpline could also be provided. Health professionals will also be in position to prescribe NRT or other treatments (for example: Varenicline or Bupropion) which can help with smoking cessation, according to routine practice. The health professional could also give advice on e-cigarette use if he or she finds it suitable.
  Arms: Standard Care

SUMMARY:
- Objective:

Our study aims to evaluate the effectiveness of the "STOP" (Sevrage Tabagique à l'aide d'Outils dédiés selon la Préférence: Smoking Cessation using preference-based tools) intervention, a preference-based smoking cessation intervention for smokers with low socio-economic position (SEP).

- Methods :

STOP is a randomised, multi-centre, single blinded, intent-to-treat trial. Participating centres include primary care practices (community, municipal or general health clinics), hospital-based facilities, and healthcare institutions specialised in addiction treatment. Smokers with low SEP will be randomised into either the intervention or control group.

Persons randomised to the control group will be accompanied by their health professional according to standard practice.

Participants randomised to the intervention group will receive the same smoking cessation advice, drug (varenicline, champix,..) prescription and support as participants in the control group, but they will also have a choice of being given free Nicotine Replacement Therapy (NRT) (transdermal patch, gum, spray, inhaler, sublingual tablets/lozenges) and/or an electronic cigarette + e-liquid on the spot to aid their quit attempt.

Follow-up appointments will take place at around 7 to 14 days, 1 month, 3 months and 6 months after inclusion, according to the participant and health professional availability.

The main outcome measure of this study will be the 7-day point prevalence tobacco abstinence at 6 months after inclusion (yes/no), defined as self-reported abstinence for at least 7 days, This self-reported abstinence will be validated by measured exhaled carbon monoxide, unless this measurement is unavailable due to the ongoing covid-19 pandemic.

DETAILED DESCRIPTION:
This is a randomised, multi-centre, single blinded, intent-to-treat pragmatic trial.

- Recruitment:

Participants will be recruited by physicians in the different study centres starting March 2021. Physicians are therefore asked to present the study to their patients who might be eligible to participate in the study. Posters and flyers inviting smokers who wish to quit to talk to their physician about smoking cessation are also supplied to participating centres.

Physicians can also carry out a pre-inclusion questionnaire over the phone or during a remote consultation, prior to a face to face appointment. However study presentation, recruitment, and baseline measures are will only be done with patients physically present at the study centre.

In some centres (depending on declared need), a research assistant (RA) might help physicians in describing the project to each potential participant. After a presentation of the study objective, a written informed consent (supplementary material) will be asked from eligible patients before proceeding with randomisation.

Recruitment period in each centre will last for up to one year, while each participant will be followed for 6 months. However, not all centers will begin recruiting at the same time, and data collection is therefore expected to last until the end of year 2023.

- Intervention standardisation: training of medical doctors:

All participating teams (investigators) will receive individual training sessions, during which we will present to them the study protocol, the randomisation procedure and the data entry (eCRF) software.

The study protocol as well as a brief reminder of recommendations concerning the use of NRT and e-cigarettes will be presented to all participating team members.

A printed study booklet summarising the study protocol will be given out to investigators as well as a digital version on a provided tablet, as well as a video format of the training session.

Further, the fidelity of the intervention will also be assured by the structured eCRF throughout the study. The eCRF will automatically determine if participants are eligible, and will guide investigators during the intervention process.

- Randomisation and blinding:

Each medical doctor (investigator) will be provided with a tablet with access to a web-based randomisation module and an Electronic Case Report Form interface (eCRF). The Randomisation will be investigator-stratified. This software is supplied by a company specialised in clinical research and will be in accordance with the latest European and French regulations regarding the protection of personal data.

After a verification of inclusion criteria, and informed consent, the module will randomise the participant either to the intervention or to the control group (1:1), and will simultaneously notify the coordinator of the study by e-mail. In order to minimise selection bias, no substitution or change of group will be permitted.

Participants will be blinded to their randomisation group: participants will not know that those randomised in the intervention group will receive free e-cigarettes and/or NRT. However, all participants - as part of the informed consent statement and the study presentation - will be informed that investigators are studying how to help smokers with their quit attempts.

Physicians - who will carry out the intervention and most of the follow up assessments - will not be blinded to treatment randomisation.

- The control group (standard care):

Participants randomised to the control group will be given standard care in assisting their smoking cessation attempt, but without free access to NRT or e-cigarettes. Standard care depends on each health professional habitual practice, it includes motivational interviewing, advice to quit and prescription of NRTs. Health professionals will also be in position to prescribe other treatments (for example: Varenicline which is covered at 65% by the French health universal insurance and might be completely covered by an additional complementary health insurance - or Bupropion which has to be paid completely). An investigator could also give advice on e-cigarette use if he or she finds it suitable.

At the end of the follow-up, participants randomised to the control group will be offered an e-cigarette + e-liquid and/or NRT in sufficient quantity for one month, if needed and desired.

- The intervention:

During the face to face baseline appointment, participants randomised to the intervention group will receive the same routine care smoking cessation advice, drug prescription and support as participants in the control group. Further, participants will also have a choice of being given free NRT (transdermal patch, gum, spray, inhaler, and sublingual tablets/lozenges) and/or e-cigarettes on the spot to aid with their quit attempt. E-cigarettes would be provided with e-liquids with different nicotine levels (3, 6, 12 and 16 mg/ml), and different flavours (tobacco, mint, and fruit).

The provided e-cigarette is the "Zlide Tube" (Shenzhen Innokin Technology Co., Shenzhen, China) an easy to use e-cigarette with a 3000mAh rechargeable battery, a 4 mL tank with sliding top refill system, provided with several spare coils, and a wall charger.

A brief and clear description of each smoking cessation aid will be given to each participant, and depending on his/her choice. At each appointment (baseline and subsequent follow-up) depending on his/her choice, he/she will be provided with a sufficient quantity to last until the following appointment. The intervention process will be guided by the eCRF which will remind investigators to list all available products, and ask them to fill the type and quantity of the delivered tools for participants in the intervention group.

Short didactic videos explaining how to use different NRTs and e-cigarettes will be available for participants in the intervention group (a mobile-friendly link to the video will be given), as well as for physicians accompanying participants.

During follow-up, participants in the intervention group can also be given other smoking cessation tools than the one(s) previously delivered, according to their preference and after seeing their physician (they can be given NRTs at the second appointment if they initially chose e-cigarette only and vice versa, or the type of given NRTs can be changed or they can receive NRT in addition to an e-cigarette). Follow-up measures after the first (baseline) appointment might take place remotely, if the participants do not require any delivery of smoking cessation tools.

Each participant in both groups will be given a diary or a "calendar postcard" on which he/she will document daily use of any smoking cessation aids, and the number of cigarettes smoked every day.

These postcards will be pre-paid and pre-addressed to return to the study investigators who would automatically fill in the corresponding data in the centralised data system.

ELIGIBILITY:
Inclusion Criteria:

* Daily smokers (5≥ cigarettes/day)
* A low socio-economic position (meaning being unemployed or being a recipient of one of the state programs for low income individuals)
* Being available for at least 4 appointments over a 6 month period
* Affiliation to or benefiting from social security or state medical support

Exclusion Criteria:

* Individuals who do not speak French, or who have cognitive impairments making it impossible to understand study information or a condition that makes it impossible for them to give informed consent.
* Major citizens protected by law, adults unable to express their consent and subject to a protective measure (guardianship, curatorship, safeguard of justice)
* Pregnant women or with a pregnancy project, mothers breastfeeding their child(ren).
* Regular smokers who vape daily (at least once a day).
* People who at the time of inclusion are already being managed for smoking cessation (whatever treatment: varenicline, electronic cigarette, NRT, hypnosis, acupuncture, psychotherapy, talk groups, etc.).
* Patients who are already participating in another clinical study (self-reported).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence at 6 months after inclusion (yes/no) | 6 months after inclusion
  Self-reported 7-day point prevalence tobacco abstinence, validated by measured exhaled carbon monoxide, if this measurement is available (depending on the sanitary measures in place due to the ongoing covid-19 pandemic).

SECONDARY OUTCOMES:
Total number of days of abstinence at 6 months | 6 months after inclusion
  Self-reported number of days without any puff
Smoking abstinence at 1 and 3 months after inclusion (yes/no) | 1 and 3 months after inclusion
  Self-reported 7-day point prevalence tobacco abstinence, validated by measured exhaled carbon monoxide, if this measurement is available (depending on the sanitary measures in place due to the ongoing covid-19 pandemic)
Number of relapses | 3 and 6 months after inclusion
  Self-reported
The number of cigarettes smoked per day | 6 months after inclusion
  Self-reported
Proportion of participants who have significantly reduced daily smoking | 6 months after inclusion
  Defined as a reduction in consumption by at least 50% in terms of the number of cigarettes smoked per day or the weight of roll-your-own tobacco per day

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHI Aix Pertuis, Aix-en-Provence
  - CHU Angers, Angers
  - Hôpital Avicenne, Bobigny
  - Hôpital Jean Verdier, Bondy
  - CH Le Vinatier, Bron
  - HCL Est, Bron
  - Hôpital Antoine Béclère, Clamart
  - Institut Coeur Poumon - Lille, Lille
  - Centre Municipal de Santé Savattero&Centre Municipal Daniel Renoult, Montreuil
  - Association Addictions France, Nîmes
  - Centre Hospitalier Sainte Anne, Paris
  - Hôpital Tenon, Paris
  - HCL Sud, Pierre-Bénite
  - Centre de Santé Pierre-Rouquès, Villejuif
  - HCL Centre, Villeurbanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Khoury F, El Aarbaoui T, Heron M, Hejblum G, Metadieu B, Le Faou AL, Ibanez G, Melchior M. Smoking cessation using preference-based tools among socially disadvantaged smokers: study protocol for a pragmatic, multicentre randomised controlled trial. BMJ Open. 2021 Jun 30;11(6):e048859. doi: 10.1136/bmjopen-2021-048859. PMID 34193499